CLINICAL TRIAL: NCT01203345
Title: Randomized Clinical Trial of Intravenous Immune Globulin (IVIG) to Prevent Neonatal Infection in Very-Low-Birth-Weight Infants
Brief Title: Intravenous Immune Globulin (IVIG) to Prevent Neonatal Infection
Acronym: IVIG
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Responsible Party: Avroy A. Fanaroff, Lead Principal Investigator, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NICHD-NRN-0002; U10HD021364 (NIH); U10HD021415 (NIH); U01HD019897 (NIH); U10HD021385 (NIH); U10HD021397 (NIH); U10HD021373 (NIH)
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2010-09

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Sepsis
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Prematurity; Septicemia; Meningitis; Urinary tract infection; Immune globulin
MeSH Terms: conditions — Premature Birth; Sepsis; Meningitis; Urinary Tract Infections | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immune globulin (Active Comparator): Lyophilized human immune globulin product
  Interventions: Drug: IVIG
- Albumin solution (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IVIG — The infants received their first dose of study drug within 24 hours of randomization.
  Other Names: Sandoglobulin
  Arms: Immune globulin
Drug: Placebo — An equal volume of 5 percent albumin solution
  Arms: Albumin solution

SUMMARY:
A controlled clinical trial was conducted at eight participating centers between January 1, 1988, and March 31, 1991. Patients were randomly assigned to an intravenous immune globulin group or a control group. There were two phases to the study (see below). During phase 1 the control infants received infusions of placebo. During phase 2 the control infants received no infusion therapy.

DETAILED DESCRIPTION:
Although survival rates for very-low-birth-weight infants (≤ 1.5 kg) continue to increase, nosocomial infections remain a major cause of morbidity and mortality. Prolonged hospitalization with exposure to resistant organisms and multiple invasive procedures, in the presence of immunologic immaturity, renders these infants vulnerable to hospital-acquired infections. Prior studies testing the ability of intravenous immune globulin to prevent nosocomial infections in premature infants have varied in design and sample size. Despite differences in the rates of observed infection, immune globulin preparations, doses, and infusion intervals, a meta-analysis of published reports suggests that nosocomial infections may be diminished by the prophylactic infusion of IgG.

The National Institute of Child Health and Human Development (NICHD) Neonatal Research Network therefore performed a prospective, multicenter, randomized trial at eight participating centers to test the hypothesis that the intravenous administration of immune globulin to infants with birth weights between 501 and 1500g would reduce the incidence of nosocomial infections.

Patients were randomly assigned to an intravenous immune globulin group or a control group. During phase 1 the control infants received infusions of placebo. During phase 2 the control infants received no infusion therapy.

ELIGIBILITY:
Inclusion Criteria:

* All neonates with birth weights of 501 to 1500 g

Exclusion Criteria:

* More than 72 hours old
* One of three or more fetuses from a multiple pregnancy
* Had infections associated with toxoplasma, rubella, cytomegalovirus, and herpes simplex viruses (the TORCH complex)
* Has a major congenital malformation, an identifiable syndrome, or a chromosomal abnormality
* Were considered nonviable
* Parental consent could not be obtained

Max Age: 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2416 (Actual)
Dates: Start 1988-01; Primary Completion 1991-03 (Actual); Study Completion 1991-03 (Actual)

PRIMARY OUTCOMES:
Incidence of nosocomial infection | 120 days of life
  Including septicemia, meningitis, or urinary tract infection

SECONDARY OUTCOMES:
Death | 120 Days of life
Morbidity | 120 days of life
  Duration of ventilator support, frequency of bronchopulmonary dysplasia, and duration of hospitalization
Local infections | 120 days of life
Necrotizing enterocolitis | 120 days of life
Specific complications of immune globulin or placebo infusion | 120 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Avroy A. Fanaroff, MD, Study Director — Case Western Reserve University; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee; Elizabeth C. Wright, PhD, Principal Investigator — George Washington University; Ronald L. Poland, MD, Principal Investigator — Wayne State University; Charles R. Bauer, MD, Principal Investigator — University of Miami; Jon E. Tyson, MD MPH, Principal Investigator — University of Texas; Joseph B. Philips, MD, Principal Investigator — University of Alabama at Birmingham; Jerold F. Lucey, MD, Principal Investigator — University of Vermont, Burlington
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - George Washington University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Wayne State University, Detroit, Michigan
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Result] Fanaroff AA, Korones SB, Wright LL, Verter J, Poland RL, Bauer CR, Tyson JE, Philips JB 3rd, Edwards W, Lucey JF, Catz CS, Shankaran S, Oh W. Incidence, presenting features, risk factors and significance of late onset septicemia in very low birth weight infants. The National Institute of Child Health and Human Development Neonatal Research Network. Pediatr Infect Dis J. 1998 Jul;17(7):593-8. doi: 10.1097/00006454-199807000-00004. PMID 9686724
- [Result] Fanaroff AA, Korones SB, Wright LL, Wright EC, Poland RL, Bauer CB, Tyson JE, Philips JB 3rd, Edwards W, Lucey JF, et al. A controlled trial of intravenous immune globulin to reduce nosocomial infections in very-low-birth-weight infants. National Institute of Child Health and Human Development Neonatal Research Network. N Engl J Med. 1994 Apr 21;330(16):1107-13. doi: 10.1056/NEJM199404213301602. PMID 8133853
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/